CLINICAL TRIAL: NCT06705296
Title: Deep Brain Stimulation (DBS) for the Treatment of Refractory Post-Traumatic Stress Disorder (PTSD)
Brief Title: Deep Brain Stimulation for Refractory PTSD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Neurosurgeon, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6355
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: PTSD
Keywords: PTSD; DBS; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study will consist of four (4) phases 1) Open label phase (from surgery until postoperative week 24); 2) Double-blinded "on/off" phase (from postoperative week 25 to 33); 3) Prolonged exposure therapy (from postoperative week 34to 44); 4) Closed-loop DBS (from postoperative week 45 to60).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Open label (Experimental): 1) Open label phase (from surgery until postoperative week 24)
  Interventions: Device: Open Label Deep Brain Stimulation
- Double-blinded "on/off" phase (Placebo Comparator): Double-blinded "on/off" phase (from postoperative week 25 to 33)
  Interventions: Device: Double blinded Deep Brain Stimulation
- Prolonged exposure therapy (Experimental): Prolonged exposure therapy (from postoperative week 34to 44)
  Interventions: Behavioral: Prolonged exposure therapy
- Closed-loop DBS (Experimental): Closed-loop DBS (from postoperative week 45 to 60).
  Interventions: Device: Closed loop Deep brain stimulation

INTERVENTIONS:
Device: Open Label Deep Brain Stimulation — Patients will receive open label deep brain stimulation
  Arms: Open label
Device: Double blinded Deep Brain Stimulation — Patients will receive double blinded deep brain stimulation
  Arms: Double-blinded "on/off" phase
Behavioral: Prolonged exposure therapy — Patients will receive prolonged exposure therapy
  Arms: Prolonged exposure therapy
Device: Closed loop Deep brain stimulation — Patients will receive closed loop deep brain stimulation
  Arms: Closed-loop DBS

SUMMARY:
Treatment refractory PTSD is a chronic and debilitating psychiatric disorder associated with high morbidity. Despite advances in neuroimaging, genetics, pharmacology and psychosocial interventions in the last half century, little progress has been made in altering the natural history of the condition or its outcome.

This study would be the first exploration of a surgical therapy for refractory PTSD. The subgenual cingulate plays a role in mechanisms of this disorder and has been successfully targeted with DBS for the treatment of depression

The study will proceed in three stages: pre-operative, operative and post-operative. In the pre-operative stage, consent will be obtained and patients will be scheduled for additional investigations, including neuroimaging (MRI), neuropsychological testing, psychophysiological testing, and a pre-operative assessment by the anesthesia service.

In the operative stage, patient will have a stereotactic frame attached directly to their skull. The patient will then undergo a computed tomography (CT) scan with the frame in place, followed by transport directly to the operating room. A skin incision will be made and two burr holes drilled through the skull. After target identification DBS electrodes will be inserted and fixed in place. Patients will be then immediately anesthetized (general anesthesia) for the next step of the surgery. This will involve implanting an internal pulse generator (IPG) under the collarbone and connecting it to the DBS electrodes.

During the post-operative phase, patients will return to the clinic 2 weeks after surgery.DBS programming visits will happen biweekly for three months, and monthly thereafter.

DETAILED DESCRIPTION:
Treatment refractory PTSD is a chronic and debilitating psychiatric disorder associated with high morbidity. Despite advances in neuroimaging, genetics, pharmacology and psychosocial interventions in the last half century, little progress has been made in altering the natural history of the condition or its outcome. It has further become increasingly accepted that this condition results, at least in part, from dysfunctional neuroanatomic circuits, whose activity and deviations can be detected with sophisticated neuroimaging techniques. Much progress has also been made in mapping the psychology of the illness to underlying neuroanatomic and neurophysiologic processes that drive and maintain these behaviours.

This study would be the first exploration of a surgical therapy for refractory PTSD. The subgenual cingulate plays a role in mechanisms of this disorder and has been successfully targeted with DBS for the treatment of depression (a highly incident co-morbidity in patients with treatment refractory PTSD).

There are currently no brain based, targeted therapies for treatment refractory PTSD with or without co-morbid depression (only the few patients described above). This study will be the first powered clinical trial exploring deep brain stimulation in this patient population.

This is a phase I, non-randomized, pilot trial for safety and efficacy of deep brain stimulation for PTSD. Patients who meet inclusion and exclusion criteria will be identified and recruited from the practices of Sunnybrook psychiatrists. The study will proceed in three stages: pre-operative, operative and post-operative. In the pre-operative stage, consent will be obtained and patients will be scheduled for additional investigations, including neuroimaging (MRI), neuropsychological testing, psychophysiological testing, and a pre-operative assessment by the anesthesia service. A clinical interview will be used to understand experiences of patients and a family member of each patient (i.e. parent, significant other, spouse, partner, informant, etc.). In the operative stage, patient will have a stereotactic frame attached directly to their skull. The patient will then undergo a computed tomography (CT) scan with the frame in place, followed by transport directly to the operating room. A skin incision will be made and two burr holes drilled through the skull. After target identification DBS electrodes will be inserted and fixed in place. Patients will be then immediately anesthetized (general anesthesia) for the next step of the surgery. This will involve implanting an internal pulse generator (IPG) under the collarbone and connecting it to the DBS electrodes . Once surgery is over, the patient will be woken up, extubated, and transferred to the recovery room. From there, patients will go to the to the neurosurgical ward (D5). During the post-operative phase, patients will return to the clinic 2 weeks after surgery.DBS programming visits will happen biweekly for three months, and monthly thereafter. Twenty (20) subjects will be enrolled and study duration for each patient will be of 60 weeks.

The study will consist of four (4) phases to be detailed below: 1) Open label phase (from surgery until postoperative week 24); 2) Double-blinded "on/off" phase (from postoperative week 25 to 33); 3) Prolonged exposure therapy (from postoperative week 34 to 44); 4) Closed-loop DBS (from postoperative week 45 to 60).

We believe that the scientific significance lay above all, in the development of a novel treatment alternative in the significant portion of this patient population who fail to respond to currently available treatments. The development of a therapy that targets brain structures known to play a role in this disease would be a substantial step forward in the treatment and understanding of these conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male patients between age 18-70
2. Diagnosis of posttraumatic stress disorder as defined by the Diagnostic and Statistical Manual fifth edition (DSM-5).
3. Treatment Resistance as defined by the persistence of clinical symptoms despite adequate treatment with four modalities, including a) selective serotonin reuptake inhibitors, b) cognitive behavioral therapy, c) other classes of medications and/or psychotherapy.
4. Severe forms of the disease as measured by Clinician Administered PTSD scale (CAPS) scores≥ 50.
5. A pattern of chronic stable PTSD lasting at least 1 year.
6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols.

Exclusion Criteria:

1. Any past or current evidence of psychosis or mania (patients with co-morbid depression will not be excluded from the study)
2. Active neurologic disease, such as epilepsy
3. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine.
4. Current suicidal ideation
5. Any contraindication to MRI or PET scanning
6. Likely to relocate or move out of the country during the study's duration.
7. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure.
8. Currently pregnant (as determined by history and serum HCG) or lactating; for females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by SAFTEE | Every 2 weeks until the 8 weeks mark, every 4 weeks until 6 month mark and every two months until the 2 year mark
  The primary objective is to establish the safety of deep brain stimulation in a patient population with treatment refractory PTSD using Systematic Assessment for Treatment Emergent Events
Clinician-Administered PTSD Scale for DSM-5 (CAPS) | Every 2 weeks until the 8 weeks mark, every 4 weeks until 6 month mark and every two months until the 2 year mark
  The CAPS assesses PTSD symptoms which have occurred in the past week.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | Every 2 weeks until the 8 weeks mark, every 4 weeks until 6 month mark and every two months until the 2 year mark
  The HAMD is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No